CLINICAL TRIAL: NCT01256580
Title: Pilot Study of Intravitreal Bevacizumab vs. Combination Therapy for Choroidal Neovascularization Secondary to Causes Other Than Age-related Macular Degeneration
Brief Title: Intravitreal Bevacizumab vs.Combination Therapy for CNV Due to Other Than AMD
Acronym: CNV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of eligible subjects.
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-10-101
Record Dates: First submitted 2010-10-29; First posted 2010-12-08 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Choroidal Neovascularization; Myopia; Punctate Inner Choroidopathy (PIC); Multifocal Choroiditis; Ocular Histoplasmosis Syndrome; Central Serous Chorioretinopathy (CSC); Angioid Streaks; Trauma, or Hereditary Eye Diseases
MeSH Terms: conditions — Choroidal Neovascularization; Myopia; White Dot Syndromes; Multifocal Choroiditis; Central Serous Chorioretinopathy; Angioid Streaks; Wounds and Injuries; Eye Diseases, Hereditary | interventions — Bevacizumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monotherapy (Active Comparator): Bevacizumab (Avastin; Genentech, Inc.)1.25 mg by intravitreal injection on day 0 and then prn (as-needed) based on ophthalmic examination and OCT findings
  Interventions: Drug: Bevacizumab (Avastin; Genentech, Inc.)
- Combination therapy (Active Comparator): Intravitreal injection of bevacizumab 1.25 mg (Avastin; Genentech, Inc.) combined with reduced fluence PDT(Visudyne®; Novartis,) and 200 ug of intravitreal dexamethasone(4mg/ml, American regent, Inc) on Day 0 and then monthly retreatment with bevacizumab as-needed and triple therapy every 3 months as-needed.
  Interventions: Drug: Bevacizumab, Dexamethasone, Verteporfin Photodynamic Therapy

INTERVENTIONS:
Drug: Bevacizumab (Avastin; Genentech, Inc.) — 1.25 mg bevacizumab (Avastin; Genentech, Inc.) by intravitreal injection
  Arms: Monotherapy
Drug: Bevacizumab, Dexamethasone, Verteporfin Photodynamic Therapy — Intravitreal injection of 1.25 mg bevacizumab (Avastin; Genentech, Inc.) combined with reduced-fluence verteporfin PDT (Visudyne®; Novartis) and 200ug of intravitreal dexamethasone
  Arms: Combination therapy

SUMMARY:
Anti-VEGF therapy has been proven efficacious for the wet (neovascular) form of macular degeneration and may be beneficial for the treatment of choroidal neovascularization (CNV) due to other causes. The limitation of this type of treatment is the necessity for frequent intraocular injections. The purpose of this study is to determine if using anti-VEGF therapy in combination with photodynamic therapy can reduce the number of treatments needed with monotherapy while achieving similar visual results. There are ongoing multicenter trials evaluating combination therapy in patients with wet AMD but no similar trial for patients with CNV due to non-AMD causes. Therefore, in this study the investigators will focus on patients with CNV not due to AMD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age > 18 years
* Clinical diagnosis of choroidal neovascularization secondary to the following causes: ocular histoplasmosis, toxoplasmosis, idiopathic, angioid streaks, choroidal ruptures, intraocular inflammation (without signs of active uveitis i.e. multifocal choroiditis), central serous retinopathy and pathologic Myopia.

Only one eye will be assessed in the study. If both eyes are eligible, the investigator and patient will determine which eye is to be treated, considering such factors as disease duration, and likelihood of response to treatment.

* Clear media and dilation to permit good stereo fundus photography
* Evidence of active CNV present on OCT images manifest by subretinal fluid, intraretinal fluid or retinal thickening ≥ 250 µm
* Best corrected VA in the study eye must be 20/40 and to 20/400 at 4 meters using ETDRS protocol.

Exclusion Criteria:

Pregnancy or lactation

* Premenopausal women not using adequate contraception The following are considered effective means of contraception: surgical sterilization; use of oral contraceptives; barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel; and IUD; or contraceptive hormone implant or patch.
* CNV secondary to AMD
* Diabetic Retinopathy
* Prior enrollment in clinical studies in the study eye
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Previous participation in another simultaneous medical investigation or trial within 1 month preceding Day 0 (excluding vitamins and minerals)
* Use of drug or treatment related or unrelated to their condition within 30 days prior to enrollment (Verteporfin, pegaptanib, ranibizumab, bevacizumab, triamcinilone or other AMD therapy in study eye)
* Concurrent use of systemic anti-VEGF therapy
* Any other ocular condition the investigator believes would pose a significant hazard to the subject if investigational treatment were initiated
* History of allergy to fluorescein
* Inability to obtain fundus photographs or FAs of sufficient quality to document CNV
* Inability to comply with study or follow-up procedures
* History of other disease, metabolic dysfunction, physical examination finding or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications.
* Current treatment for active systemic infection
* History of uncontrolled glaucoma (defined as intraocular pressure >30mmHg despite treatment with anti-glaucoma medication) or filtering surgery in the study eye
* Family history of glaucoma
* Patients who have undergone intraocular surgery within last 2 months
* Aphakia or absence of the posterior capsule in the study eye Previous violation of the posterior capsule in the study eye is also excluded unless it occurred as a result of YAG posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Mean number of treatments per group | 12 months

SECONDARY OUTCOMES:
Mean change in visual acuity from baseline | 12 months
  Mean change in visual acuity from baseline
  * Proportion of subjects losing ≤8 letters (≈1.5 lines) from baseline
  * Proportion gaining ≥15 letters from baseline
  * Proportion with a Snellen equivalent of 20/200 or worse (legal blindness = 20/200 or worse in both eyes)
  * Mean change from baseline in total area of CNV and total area of leakage from CNV from baseline to month 12 by FA Mean change in central subfield macular thickness (CMT) measured by OCT from baseline to month 12 Change of in areas of hypoautofluorescence (indicating atrophy) from baseline to month 12

CONTACTS AND LOCATIONS:
Overall Officials: Ivana K Kim, MD, Principal Investigator — Massachussetts Eye& Ear Infirmary

REFERENCES:
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203